CLINICAL TRIAL: NCT05637385
Title: Training Oculo-motor Control to Improve Vision When Using a Preferred Retinal Locus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Russell L. Woods (Other)
Collaborators: Research to Prevent Blindness / Lions Club International Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Russell L. Woods, Associate Scientist, Schepens Eye Research Institute
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P002309
Record Dates: First submitted 2022-11-04; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Central Visual Impairment
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Intervention Model Description: Two-way mixed (one within, one between) factor study. Same training, applied to central vision loss group and normal vision control group viewing with simulated central scotomas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- central vision loss (Experimental): will receive behavioral intervention
  Interventions: Behavioral: Training of perception and oculo-motor control
- normal vision (Active Comparator): using simulated central scotomas, will receive behavioral intervention
  Interventions: Behavioral: Training of perception and oculo-motor control

INTERVENTIONS:
Behavioral: Training of perception and oculo-motor control — Behavioral training of eye movements and perception

SUMMARY:
When high-detail vision is lost due to a retinal disease such as macular degeneration, people see poorly, and have difficulty with eye movements (oculo-motor control). This preliminary study will investigate a potential behavioral intervention that may improve the ability to perform vision-related daily activities such as reading, recognising faces and watching television. The intervention involves many sessions that will train visual perception and eye movements over a period of a few months. Participants will have either lost central vision in both eyes or have normal vision (control group).

DETAILED DESCRIPTION:
The purpose of the study is evaluate a potential treatment for loss of (foveal) central vision in both eyes which results in the use of a preferred retinal locus (PRL). The treatment is a series of 16 sessions of about one-hour duration that will involve a mixture of oculomotor control (OMC) training, perceptual training, and scotoma awareness. Two groups will receive the training: (1) central vision loss; and (2) normal sight who will use a simulated scotoma (called control group below).

A single-site, two-way mixed factor, one within-subject and one between-subject, minimal-risk phase-2 study. Each participant with vision loss or in the control group will attend for three outcome-measurement visits and 16 training visits over a period of about two months (at 2 visits per week). Feasibility metrics will be obtained during recruitment and study conduct. PRL and OMC metrics will be obtained at every visit. Outcome metrics will be obtained before treatment, following 8 training sessions, and following 16 training sessions.

Participants in the control group will experience a simulated central scotoma created by a gaze-contingent visual display system that simulates the loss of central vision by obscuring a region of central vision during testing and training.

Participants will be trained using an integrated oculo-motor and perceptual training approach using a gaze-contingent visual display to provide scotoma awareness. Two tasks will alternate: (1) a textured search target that suddenly shifts, drifts smoothly, or is stable, requiring the subject to make a saccade, a smooth pursuit, or fixate, respectively, following which there is a same-different task to test attention; and (2) target following and visual search for (a) face within distractors, (b) object recognition and location, and (c) word recognition and object identification over cluttered background. During training, for the vision-loss group, the binocular scotoma (created by the retinal lesions) will be outlined using a gaze-contingent system, so that the subject will see a border at the edge of their binocular scotoma that moves with gaze, alerting them to the location of the scotoma.

In addition to the 16 training sessions, there will be longer (2.5 to 3 hours) measurement sessions: (1) before training; (2) after 8 training sessions; and (3) after 16 training sessions. Due to the number of procedures, the first measurement session might consist of two sessions. Thus, each participant with vision loss will participate in 19 or 20 sessions in total.

Ideally, participants will attend for two visits per week. However, the schedule is flexible and can be adapted to a participants schedule.

ELIGIBILITY:
Central Vision Loss Group

Inclusion Criteria:

* Bilateral foveal loss that includes the fovea in each eye, as determined through retinal examination
* fluent in English
* Cognitive function MoCA (Montreal Cognitive Assessment) test >20
* Binocular visual acuity 20/800 or better
* able to sit for at least an hour

Exclusion Criteria:

* speech impediment
* history of neurological or psychiatric disease
* inability to provide informed consent
* inability to follow instructions in English

Normal Vision Control Group

Inclusion Criteria:

* fluent in English
* Cognitive function MoCA (Montreal Cognitive Assessment) test >25
* Binocular visual acuity 20/40 or better
* able to sit for at least an hour

Exclusion Criteria:

* any ophthalmic disease that might impact on the conduct of the study, especially conditions that cause vision field loss
* speech impediment
* history of neurological or psychiatric disease
* inability to provide informed consent
* inability to follow instructions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
reading speed following eight training sessions | comparing reading speed before intervention and after 8 sessions of training
  reading of paragraphs of text
reading speed following sixteen training sessions | comparing reading speed before intervention and after 16 sessions of training
  reading of paragraphs of text
face discrimination threshold following eight training sessions | comparing face discrimination thresholds before intervention and after 8 sessions of training
  recognizing differences between faces
face discrimination threshold following sixteen training sessions | comparing face discrimination thresholds before intervention and after 16 sessions of training
  recognizing differences between faces
video comprehension (shared word score) following eight training sessions | comparing shared word scores before intervention and after 8 sessions of training
  understanding and describing the content of short video clips
video comprehension (shared word score) following sixteen training sessions | comparing shared word scores before intervention and after 16 sessions of training
  understanding and describing the content of short video clips

SECONDARY OUTCOMES:
PRL location relative to the location before the intervention (training) | location at each of the 16 training sessions as compared to the location before intervention
  location of the preferred retinal locus measured from a retinal image obtained during a fixation examination
Oculo-motor reference location relative to the location before the intervention (training) | at each of the 16 training sessions as compared to the location before intervention
  first landing location of saccades to a new location measured using a gaze tracking system; measures whether there has been an adjustment of eye movement planning
saccade dynamics relative to the location before the intervention (training) | at each of the 16 training sessions as compared to the location before intervention
  slope of the saccadic main sequence, which is the speed to distance relationship of saccades (fast eye movements), as measured using a gaze tracking system
single-letter visual acuity following eight training sessions | comparing visual acuity before intervention and after 8 sessions of training
  ability to read single letters of varying size
single-letter visual acuity following sixteen training sessions | comparing visual acuity before intervention and after 16 sessions of training
  ability to read single letters of varying size
letter contrast sensitivity following eight training sessions | comparing letter contrast sensitivity before intervention and after 8 sessions of training
  ability to read "large" letters of low contrast
letter contrast sensitivity following sixteen training sessions | comparing letter contrast sensitivity before intervention and after 16 sessions of training
  ability to read "large" letters of low contrast
Geriatric Depression Scale (GDS) following eight training sessions | comparing GDS scores before intervention and after 8 sessions of training
  evaluate depression and aspects of quality of life
Geriatric Depression Scale (GDS) following sixteen training sessions | comparing GDS scores before intervention and after 16 sessions of training
  evaluate depression and aspects of quality of life
Veterans Affairs Low Vision Visual Functioning Questionnaire (VA LV VFQ) following eight training sessions | comparing VA LV VFQ scores before intervention and after 8 sessions of training
  measure of visual ability and vision-related limitations
Veterans Affairs Low Vision Visual Functioning Questionnaire (VA LV VFQ) following sixteen training sessions | comparing VA LV VFQ scores before intervention and after 16 sessions of training
  measure of visual ability and vision-related limitations

OTHER OUTCOMES:
enrollment rate | duration of enrollment period
  compares the number of participants who enroll in the study to the number of potential participants identified; and the time taken to enroll the study sample, and reasons for lack of willingness to participate (qualitative)
retention rate | duration of intervention period
  compares the number of participants who complete the study to the number of participants who enrolled in the study; and obtain reasons for dropout
treatment fidelity | duration of intervention period
  adherence to the treatment session schedule, the adherence rate, any adherence pattern, and reasons for adherence failures
measurement fidelity | duration of intervention period
  ability to obtain outcome measures (proportion of outcome measures completed, period and variance of improvement across subjects), obtain feedback on acceptability of outcome measures, and qualitative reasons for failure to complete specific outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Russell L Woods, PhD, Principal Investigator — Schepens Eye Research Institute

IPD SHARING:
Plan to Share IPD: Undecided
If approved by our IRB (Institutional Review Board), we may be able to share de-identified outcome metrics and eye movement measurements. A data use agreement would be required.